CLINICAL TRIAL: NCT03016845
Title: Pharmacokinetics of Ciprofloxacin in Critically Ill Patients - a Screening Study to Assess the Feasibility of Renal Function Markers to Predict Ciprofloxacin Clearance (CAPOEIRA)
Brief Title: Pharmacokinetics of Ciprofloxacin in Critically Ill Patients
Acronym: CAPOEIRA
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Canisius-Wilhelmina Hospital (Other); UMC Utrecht (Other); Gelderse Vallei Hospital (Other); Tergooi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UMCN-AFK 16.07
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2017-11

CONDITIONS: Bacterial Infections
Keywords: ciprofloxacin; pharmacokinetics; Intensive Care Unit; Cystatin C; CKD-EPI; renal function
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma samples for determination of ciprofloxacin and cystatin C Urine for measuring 24h creatinine cleaurance
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Optimal understanding of ciprofloxacin pharmacokinetics in critically ill patients is lacking resulting in large variation of achieved exposure and possible inadequate therapy. The investigators hypothesize that drug dosing based on CKD-EPIcr-cys provides a useful method to individualize and optimize therapy for ciprofloxacin and eventually improve outcome.

In a multi-centre, observational, open-label study the investigators aim to define : the model for estimation of renal function that most accurately predicts ciprofloxacin clearance in critically ill patients.

DETAILED DESCRIPTION:
Correct estimation of glomerular filtration rate (GFR) is necessary in critically ill patients in order to asses renal function. GFR is subsequently used to derive and appropriate drug dosing of renally excreted drugs and warrant adequate dose adaptations.

It is known that estimation of GFR based on creatinine clearance is not precise, especially in populations with altered muscle mass or instable renal function, such as the Intensive Care Unit (ICU) population.

The use of combined filtration markers together, cystatin C and creatinine, can improve precision in estimating GFR (eGFR). Studies confirmed that eGFR based on both creatinine and cystatin C is more precise than eGFR creatinine or eGFR cystatin C. The equation based on both creatinine and cystatin C, the Chronic Kidney Disease Epidemiology Collaboration creatinine-cystatin C (CKD-EPIcr-cys), may therefore improve eGFR and thus drug dosing in ICU patients, a population that does not reach PK/PD targets frequently.

So far little is known about drug dosing based on CKD-EPIcr-cys. Currently optimal understanding of ciprofloxacin pharmacokinetics in critically ill patients is lacking, resulting in large variation of achieved exposure and possible inadequate therapy. The investigators hypothesize that drug dosing based on CKD-EPIcr-cys provides a useful method to individualize and optimize therapy for ciprofloxacin and eventually improve outcome.

In a multi-centre, observational, open-label study the investigators aim to define the model for estimation of renal function that most accurately predicts ciprofloxacin clearance in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is admitted to an ICU
2. Subject is at least 18 years on the day of the first dosing
3. Is managed with an arterial line or central venous catheter
4. Is managed with an urinary catheter
5. Is already treated with ciprofloxacin as part of routine clinical care

Exclusion Criteria:

1. Has previously participated in this study
2. Is on renal replacement therapy (RRT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving ciprofloxacin for treating a suspected or proven bacterial infection at the ICU will be included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
model for estimation of renal function that most accurately predicts ciprofloxacin clearance | Day 1 and day 2
  Full pharmacokinetic curves will be taken on Day 1 and Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Roger Bruggemann, Principal Investigator — Radboud University Medical Center
Locations (4):
- Netherlands (4):
  - Ziekenhuis Gelderse Vallei, Ede
  - CWZ, Nijmegen
  - Radboudumc, Nijmegen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gieling EM, Wallenburg E, Frenzel T, de Lange DW, Schouten JA, Ten Oever J, Kolwijck E, Burger DM, Pickkers P, Ter Heine R, Bruggemann RJM. Higher Dosage of Ciprofloxacin Necessary in Critically Ill Patients: A New Dosing Algorithm Based on Renal Function and Pathogen Susceptibility. Clin Pharmacol Ther. 2020 Oct;108(4):770-774. doi: 10.1002/cpt.1855. Epub 2020 May 15. PMID 32298468
- See also: paper — https://pubmed.ncbi.nlm.nih.gov/32298468/